CLINICAL TRIAL: NCT02374957
Title: Cilostazol After Lower Extremity Arterial Revascularization Trial (CLEAR)
Brief Title: Cilostazol After Lower Extremity Arterial Revascularization Trial
Acronym: CLEAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Original PI left institution
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00030275
Record Dates: First submitted 2015-02-10; First posted 2015-03-02 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Peripheral Arterial Disease; Claudication (Finding)
Keywords: leg pain; claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Signs and Symptoms | interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cilostazol (Active Comparator): Administer Cilostazol100 mg twice daily for 90 days.
  Interventions: Drug: Cilostazol
- Control (No Intervention): No Cilostazol

INTERVENTIONS:
Drug: Cilostazol — 100 mg twice daily for 90 days
  Other Names: Pletal
  Arms: Cilostazol

SUMMARY:
Twenty patients will be recruited to CLEAR. Ten will be randomized to the treatment arm (Cilostazol) and tenwill be randomized to the control group. Patients randomized to the treatment arm will receive Cilostazol for 90 days. The primary purpose of this study is to collect quality of life data on patients undergoing peripheral revascularization in order to determine the sample size required to adequately power a trial of Cilostazol versus usual care without Cilostazol and its effect on quality of life.

DETAILED DESCRIPTION:
Cilostazol is the only medication approved for use in peripheral arterial disease (PAD) patients to reduce claudication symptoms. Contemporary data has demonstrated that Cilostazol improves patency after endovascular interventions in multiple randomized trials and retrospective studies done in Japan in both critical limb ischemia and claudication patients. However, Cilostazol use after peripheral revascularization has been sporadic and there has been no research to estimate patient quality of life with use of Cilostazol after open or endovascular lower extremity revascularization.

This is a prospective investigator initiated single-center open-label, non-placebo controlled pilot study. Eligible patients would be randomized to either the Cilostazol treatment or the non-Cilostazol treatment groups using a closed envelope randomization technique. Twenty patients will be recruited and randomized; Ten to the treatment group and tento the control group.

The primary purpose of this pilot study is to collect quality of life data on patients undergoing peripheral revascularization in order to determine the sample size required for adequate powered trial of Cilostazol versus usual care without Cilostazol and its effect on Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* At least 35 years of age
* Atherosclerotic peripheral arterial disease
* Able to provide informed consent
* Lower extremity open or endovascular revascularization.

Exclusion Criteria:

* Known CHF (class III/IV)
* Allergic reaction to phosphodiasterase inhibitors
* Intracranial bleeding within 3 months or active bleeding peptic ulcer disease
* Traumatic vascular injuries requiring revascularization
* Pregnant or breast feeding women or women who plan to get pregnant over the study period
* Planned ipsilateral major amputation within 30 days of index procedure
* Moderate to severe hepatic impairment.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Edwards, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cilostazol | Control
Started | 11 | 9
Completed | 10 | 9
Not Completed | 1 | 0
Not completed — Patient did not complete forms correctly | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilostazol | Control | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 63.60 [52 to 82] | 63.11 [43 to 73] | 63.37 [43 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life in Relation to Use of Cilostazol After Lower Extremity Revascularization (EQ-5D Sum Score) at 6 Weeks
Description: The Euroqol 5D (EQ5D) questionnaire will be completed at baseline, six weeks and three months follow-up. Cross-sectional and change scores will be used to project sample size requirements for a full trial. The EuroQol (EQ-5D) questionnaire is a standardized instrument for measuring generic health status. The descriptive system consists of the following five dimensions: 1) mobility, 2) self-care, 3) usual activities, 4) pain/discomfort, 5 anxiety/depression. Each participant was asked to choose one level that reflects their own health state today for each of the five dimensions. The EQ5D sum score is a composite sum of the individual dimension scores. Values of the total score can range from 5 to 25 with higher scores indicating a worse health state. Separate change scores are estimated at each follow-up time point.
Time Frame: Baseline and 6 weeks.
Population: Only patients with data collected at each pair of time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 9 | 7
score on a scale
  Baseline | 14.00 (4.00) | 15.57 (2.94)
  Six Weeks | 12.89 (3.33) | 12.14 (4.53)
  Six Week Change Score | 1.11 (3.89) | 3.43 (3.95)
Statistical Analysis 1: Comparison: Cilostazol vs Control; Null hypothesis: six-week change in EQ5D sum score is the same between the two arms. Alternate hypothesis: one arm experiences more change in EQ5D than the other over initial six weeks (two-sided test); Test type: Superiority; p = 0.26, t-test, 2 sided

2. Primary Outcome: Change in Quality of Life in Relation to Use of Cilostazol After Lower Extremity Revascularization (EQ-5D Sum Score) at 3 Months
Description: The Euroqol 5D (EQ5D) questionnaire will be completed at baseline, six weeks and three months follow-up. Cross-sectional and change scores will be used to project sample size requirements for a full trial. The EuroQol (EQ-5D) questionnaire is a standardized instrument for measuring generic health status. . The descriptive system consists of the following five dimensions: 1) mobility, 2) self-care, 3) usual activities, 4) pain/discomfort, 5 anxiety/depression. Each participant was asked to choose one level that reflects their own health state today for each of the five dimensions. The EQ5D sum score is a composite sum of the individual dimension scores. Values of the total score can range from 5 to 25 with higher scores indicating a worse health state. Separate change scores are estimated at each follow-up time point.
Time Frame: Baseline and 3 months
Population: Only patients with data collected at each pair of time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline | 14.50 (4.07) | 16.17 (2.71)
  Three Months | 13.75 (4.62) | 12.50 (3.21)
  3 Month Change Score | 0.75 (3.77) | 3.67 (3.50)
Statistical Analysis 1: Comparison: Cilostazol vs Control; Null hypothesis: three-month change in EQ5D sum score is the same between the two arms. Alternate hypothesis: one arm experiences more change in EQ5D than the other over three months (two-sided test); Test type: Superiority; p = 0.17, t-test, 2 sided

3. Primary Outcome: Change in Quality of Life in Relation to Use of Cilostazol After Lower Extremity Revascularization (Euroqol-5D Visual Analog) at 6 Weeks.
Description: The Euroqol 5D (EQ5D) questionnaire will be completed at baseline, six weeks and three months follow-up. Cross-sectional and change scores will be used to project sample size requirements for a full trial. The EuroQol (EQ-5D) questionnaire is a standardized instrument for measuring generic health status. The second part of the Euroqol-5D is a analog scale with endpoints labeled "best imaginable health state" and "worst imaginable health state" with 0 representing worst health state and 100 representing best health state. Participants choose which number best represents their health on that day. Separate change scores are estimated at each follow-up time point.
  Higher numbers are better.
Time Frame: Baseline and Six Weeks
Population: Only patients with data collected at each pair of time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 9 | 7
score on a scale
  Baseline | 61.67 (17.32) | 42.86 (22.33)
  Six Weeks | 60.00 (24.37) | 71.43 (23.40)
  6 Week Change Score | -1.67 (21.94) | 28.57 (27.04)
Statistical Analysis 1: Comparison: Cilostazol vs Control; Null hypothesis: six-week change in EQ5D visual analog score is the same between the two arms. Alternate hypothesis: one arm experiences more change in EQ5D visual analog score than the other over initial six weeks (two-sided test); Test type: Superiority; p = 0.027, t-test, 2 sided

4. Primary Outcome: Change in Quality of Life in Relation to Use of Cilostazol After Lower Extremity Revascularization (Euroqol-5D Visual Analog) at 3 Months.
Description: as for outcome 3
Time Frame: Baseline and 3 months
Population: Only patients with data collected at each pair of time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline | 57.50 (13.89) | 41.67 (24.22)
  Three Months | 47.50 (21.88) | 65.83 (28.00)
  3 Month Change Score | -10.00 (14.14) | 24.17 (29.73)
Statistical Analysis 1: Comparison: Cilostazol vs Control; Null hypothesis: three-month change in EQ5D visual analog score is the same between the two arms. Alternate hypothesis: one arm experiences more change in EQ5D visual analog score than the other over three months (two-sided test); Test type: Superiority; p = 0.014, t-test, 2 sided

5. Primary Outcome: Change in Quality of Life Scores - Estimation of Ambulatory Capacity by History-Questionnaire (EACH-Q) at 6 Weeks
Description: The quality of life instrument EACH Q questionnaire was administered at baseline, 6-week and 3-month follow-up visits. Cross-sectional and change scores will be used to project sample size requirements for a full trial. The EACH-Q is a four-item questionnaire that estimates the maximum duration that patients can maintain different displacement speeds, ranging from "slow walk" to "running." Values of the total score can range from 0 to 100 with higher scores indicating a better health state. Separate change scores are estimated at each follow-up time point.
  With the EACH-Q higher scores are better.
Time Frame: Baseline and Six Weeks
Population: Only patients with data collected at each pair of time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 9 | 7
score on a scale
  Baseline | 17.11 (8.82) | 16.43 (10.91)
  Six Weeks | 13.78 (9.20) | 11.71 (7.91)
  Change Score | -3.33 (12.04) | -4.71 (11.51)
Statistical Analysis 1: Comparison: Cilostazol vs Control; Null hypothesis: six-week change in EACH Q sum score is the same between the two arms. Alternate hypothesis: one arm experiences more change in EACH Q sum score than the other over initial six weeks (two-sided test); Test type: Superiority; p = 0.82, t-test, 2 sided

6. Primary Outcome: Change in Quality of Life Scores - Estimation of Ambulatory Capacity by History-Questionnaire (EACH-Q) at 3 Months
Description: as for outcome 5
Time Frame: Baseline and 3 months
Population: Only patients with data collected at each pair of time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline | 13.38 (9.15) | 15.50 (11.64)
  Three Months | 15.25 (18.91) | 13.00 (10.94)
  3 Month Change Score | 1.88 (17.01) | -2.50 (12.83)
Statistical Analysis 1: Comparison: Cilostazol vs Control; Null hypothesis: three-month change in EACH Q sum score is the same between the two arms. Alternate hypothesis: one arm experiences more change in EACH Q sum score than the other over three months (two-sided test); Test type: Superiority; p = 0.61, t-test, 2 sided

7. Secondary Outcome: Graft Patency, Determined as Opened or Occluded by Duplex Scan Post-intervention.
Description: Graft patency was determined by duplex scan as opened or occluded. Follow-up duplex testing ranged from 13 days to 259 days. Number of patency failures (i.e., graft occlusions) are shown below by treatment arm.
Time Frame: 13 days to 259 days
Population: One patient had no scans to determine graft patency.
Measure: Count of Participants; unit: Participants
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 10 | 8
Participants | 3 | 2
Statistical Analysis 1: Comparison: Cilostazol vs Control; Null hypothesis: time to patency-failure (graft occlusion) is the same between treatment arms. Alternate hypothesis: one arm differs from the other in durability of graft patency (two-sided test); Test type: Superiority; p = 0.26, Log Rank

8. Other Pre Specified Outcome: Number of Participants Affected by Death
Description: Number of Participants affected by Death was reported
Time Frame: 90 days
Population: Overall survival
Measure: Count of Participants; unit: Participants
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 10 | 9
Participants | 0 | 1

9. Other Pre Specified Outcome: Patients Who Had Amputations Following Initial Procedure.
Description: Patients who went on to have amputations following initial procedure
Time Frame: 90 days
Population: Nineteen patients randomized to either Cilostazol or Control group who had lower extremity revascularization.
Measure: Count of Participants; unit: Participants
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 10 | 9
Participants | 1 | 2

10. Other Pre Specified Outcome: Number of Participants Who Had a Stroke
Description: Secondary outcome measure - patients who had a stroke during the 90 day follow up period.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

11. Other Pre Specified Outcome: Claudication Symptoms and Rest Pain.
Description: Secondary outcome measures including claudication symptoms and rest pain.
Time Frame: 90 days
Population: No data collected due to early termination of study.
Arm/Group | Cilostazol | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days from surgery.
Description: Adverse events include but are not limited to hospitalized CHF, MI, stroke, amputation, pneumonia.
Arm/Group | Cilostazol | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/9
Serious Adverse Events (participants affected / at risk) | 3/10 | 3/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol (N=10) | Control (N=9)
Amputation (Surgical and medical procedures) | 1 (1) | 2 (2) — Patients went on to have amputations after initial procedure.
Hemodialysis (Renal and urinary disorders) | 1 (1) | 1 (1) — Patient went on to diaysis
Other non-CVD (Renal and urinary disorders) | 1 (1) | 0 (0) — Renal Mass
Suspected MI (Cardiac disorders) | 0 (0) | 1 (1) — Patient expired from suspected myocardial infarction

LIMITATIONS AND CAVEATS:
The original principle investigator decided to terminate the study early in order to begin analysis due to his impending departure from Wake Forest Baptist Health.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT02374957/Prot_SAP_000.pdf